CLINICAL TRIAL: NCT03652493
Title: Multicentre, Open-label Phase 2 Trial Evaluating the Efficacy of CARBOPLATIN in Metastatic Prostate Cancer With Gene Alterations in the Homologous Recombination Pathway
Brief Title: Trial Evaluating the Efficacy of CARBOPLATIN in Metastatic Prostate Cancer With Gene Alterations in the Homologous Recombination Pathway
Acronym: PRO-CARBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: French Interregional Group of Clinical Research and Innovation (Other); Ligue Contre le Cancer (French association Against Cancer) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004764-35
Record Dates: First submitted 2018-07-25; First posted 2018-08-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2021-06

CONDITIONS: Castration-resistant Prostate Cancer; Metastasis
Keywords: Anomaly of the Homologous Recombination (HR) pathway; Carboplatin
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARBOPLATIN (Experimental): CARBOPLATIN in Intraveinous Dose AUC 5 according to Calvert every 3 weeks, for a duration of 6 to 9 cycles
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Tumoral evaluation every 3 cycles

SUMMARY:
The investigators propose a phase II study to evaluate the efficacy of carboplatin monotherapy in the tumor subgroup of metastatic castration-resistant prostatic carcinomas with somatic abnormality in the Homologous Recombination (HR) pathway.

This study may also better characterize the molecular abnormalities of tumors required for the carboplatin response

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Patients with adenocarcinoma or poorly differentiated prostate carcinoma, histologically confirmed (small-cell histology or high-grade neuroendocrine histology excluded)
* Tumor presenting a somatic pathogenic variant likely to alter the homologous recombination pathway previously detected on a tumor biopsy or on circulating tumor DNA, or germinal mutation among the list of genes defined in the study
* Castration-resistant tumor defined by progression despite well-conducted androgen deprivation treatment: testosterone ≤50ng /dL agonist / antagonist of luteinizing hormone-releasing hormone (LHRH) or surgical castration. The patient must agree to continue concomitant LHRH-mediated (agonist or antagonist) therapy throughout the duration of the study regimen for patients with no history of surgical castration.
* Patients must have performed at least one line of chemotherapy by taxane in case of castration resistance:

  * Patients who have received docetaxel treatment in a hormone-sensitive situation must have received at least treatment with cabazitaxel in case of castration resistance
  * Patients who have not received chemotherapy in a hormone-sensitive situation must have received docetaxel AND cabazitaxel or have a contraindication to discontinue treatment.
* Patients must have been treated with at least 2nd generation hormone therapy (eg, abiraterone acetate or enzalutamide)
* Patients may have been treated with a poly (ADP-ribose) polymerase inhibitor (PARP)
* Performance Status <2
* Metastatic disease progressive

Exclusion Criteria:

* Absence of previous treatment with taxane in situation of sensitivity or resistance to castration.
* Absence of previous treatment with cabazitaxel in case of resistance to castration (except contraindication explaining the non-administration of treatment)
* No treatment with 2nd generation hormone therapy (eg abiraterone acetate or enzalutamide) unless contraindicated to explain non-administration of treatment
* Previous treatment with platinum
* Symptomatic and untreated central nervous system (CNS) metastases. Patients with asymptomatic and pre-treated CNS metastases are included if they are clinically stable (not requiring corticosteroid therapy for 28 days) and must have a brain MRI evaluation at screening and during follow-up.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of carboplatin on metastatic prostatic carcinoma resistant to castration Efficacy of carboplatin: The best radiological tumoral response rate | Up to 27 weeks (9 cycles)
  Tumoral response rate (TR) defined according to the recommendations of the PCWG3 criteria : Objective radiological response
Efficacy of carboplatin: biological response rate defined by value of PSA | Up to 27 weeks (9 cycles)
  Biological response rate (TR) defined according to the recommendations of the PCWG3 criteria : Decrease of PSA ≥ 50%,

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Chu Rouen, Rouen
  - Institut Gustave ROUSSy IGR, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coquan E, Penel N, Lequesne J, Leman R, Lavaud P, Neviere Z, Brachet PE, Meriaux E, Carnot A, Boutrois J, Castera M, Goardon N, Muller E, Leconte A, Thiery-Vuillemin A, Clarisse B, Joly F. Carboplatin in metastatic castration-resistant prostate cancer patients with molecular alterations of the DNA damage repair pathway: the PRO-CARBO phase II trial. Ther Adv Urol. 2024 Feb 28;16:17562872241229876. doi: 10.1177/17562872241229876. eCollection 2024 Jan-Dec. PMID 38425504